CLINICAL TRIAL: NCT02724592
Title: Effect of Self Assembling Peptide P11-4 in Patients With Early Occlusal Carious Lesions: A Mono-centre, Controlled, Single-blinded, Randomised Study
Brief Title: Self Assembling Peptide P11-4 in Patients With Early Occlusal Carious Lesions
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BB001/13
Record Dates: First submitted 2016-03-07; First posted 2016-03-31 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): intervention group, self assembling peptide P11-4 (Curodont™ Repair) and fluoride varnish (Duraphat®)
  Interventions: Device: self assembling peptide P11-4 (Curodont™ Repair); Device: fluoride varnish (Duraphat®)
- control (Active Comparator): control group, only Fluoride varnish (Duraphat®)
  Interventions: Device: fluoride varnish (Duraphat®)

INTERVENTIONS:
Device: self assembling peptide P11-4 (Curodont™ Repair) — Applying of self assembling peptide P11-4 (Curodont™ Repair) on teeth with initial caries lesions
  Arms: intervention
Device: fluoride varnish (Duraphat®) — Applying fluoride varnish (Duraphat®) on teeth with initial caries lesions

SUMMARY:
Objectives: Occlusal surfaces of erupting permanent molars are highly prone to caries. Self-assembling peptide (P11-4) has proven to enhance biomimetic mineralization of early carious lesions. Aim of this study was to evaluate safety, clinical applicability and effect of using P11-4 (Curodont™ Repair) in non-invasive treatment of early occlusal lesions.

Methods: 70 patients with active early occlusal lesions (ICDAS-II:1-3) on first or second permanent molars at eruption will be allocated in this randomized, controlled, single blinded study to test (Curodont™ Repair+Duraphat®) or control (Duraphat®) groups.

DETAILED DESCRIPTION:
Objectives: Occlusal surfaces of erupting permanent molars are high prone to caries. Self-assembling peptide (P11-4) has proven to enhance biomimetic mineralization of early carious lesions. Aim of this study was to evaluate safety, clinical applicability and effect of using P11-4 (Curodont™ Repair) in non-invasive treatment of early occlusal lesions.

Methods: 70 patients with active early occlusal lesions (ICDAS-II:1-3) on first or second permanent molars at eruption will be allocated in this randomized, controlled, single blinded study to test (Curodont™ Repair+Duraphat®) or control (Duraphat®) groups. Safety and applicability will be evaluated using dentist's/patient's questionnaires about adverse events, difficulties of application and satisfaction with procedure. Lesions will be assessed at baseline and recalls after 3 and 6 months regarding caries activity, clinical status (ICDAS-II) and with Diagnodent®. The Visual Analog Scale (VAS) of regression and of lesion size in addition to the Global Impression of Change Questionnaire will also be assessed. At every recall, fluoride varnish will be applied on lesions and patients received oral health instructions.

ELIGIBILITY:
Inclusion Criteria:

* Early occlusal carious lesions (without cavity) on permanent molar "6" or "7" at eruption which does not require an invasive treatment
* Age ≥ 5 years
* Size and form of the lesions: the lesions must both be fully visible and assessable and accessible
* Willing and able to attend the on-study visits and to observe good oral hygiene throughout the study
* Written informed consent before participation in the study

Exclusion Criteria:

* Evidence of tooth erosion
* Fluoride varnish application < 3 months prior to study treatment
* History of head and neck illnesses (e.g. head/neck cancer)
* Any pathology or concomitant medication affecting salivary flow or dry mouth
* Any metabolic disorders affecting bone turnover
* Concurrent participation in another clinical trial

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Alkilzy, Dr. PhD, Principal Investigator — University of Greifswald

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alkilzy M, Tarabaih A, Santamaria RM, Splieth CH. Self-assembling Peptide P11-4 and Fluoride for Regenerating Enamel. J Dent Res. 2018 Feb;97(2):148-154. doi: 10.1177/0022034517730531. Epub 2017 Sep 11. PMID 28892645

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 70 patients met the inclusion criteria and offered participation
Pre-assignment Details: No patient declined to participate
Period: Overall Study
Arm/Group | Intervention | Control
Started | 35 | 35
Completed | 31 | 34
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Full Range); unit: years] | 9.0 [7.0 to 13.0] | 10.5 [8.0 to 13.0] | 9.75 [7.0 to 13.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 22 | 21 | 43
Region of Enrollment [Number; unit: participants]
  Germany | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Caries Activity and Progression Assessment Using LASER Fluorescence Readings by Diagnodent® Device.
Description: Evaluation of the additional therapeutic benefit of Curodont™ compared to fluoride varnish (Duraphat®) alone on early occlusal carious lesions using LASER "Light Amplification by Stimulated Emission of Radiation" fluorescence readings by Diagnodent® device.
  Diagnodent® device measures the caries activity using LASER fluorescence of bacterial secretions in the caries lesion. The readings range from 0 to 99; 0 means no bacterial activity in the carious lesion whereas 99 refers to high bacterial and caries activity.
  Effect via the changes in LASER fluorescence readings between Baseline and 6-months recall (Change = Baseline value - 6 months value). Higher positive change value means caries regression, whereas lower positive or negative change value refers to caries progression.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 31 | 34
units on a scale | 18.6 (19.8) | 1.1 (25.8)

2. Secondary Outcome: Visual Analog Scale of Lesion Progression (VAS)
Description: Visual Analog Scale of lesion progression (VAS), Effect via t test between Baseline and 6-months recall VAS values range from -100 % to +100 %. The value of -100 means that the carious lesion is strongly remineralising, the value of 0 means that the lesion is arrested, and the value of +100 means that the lesion is strongly progressing.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 31 | 34
units on a scale | 88.0 (40.8) | 49.1 (43.8)

3. Secondary Outcome: ICDAS Classification Index
Description: Number of patients who have improvement on the ICDAS classification index (International Caries Detection and Assessment System), changes from Baseline to 6-months recall.
  This carries clinical index range from 0 to 6. The values mean:
  0 No evidence of caries
  1. Initial caries
  2. Distinct visual change in enamel
  3. Localised enamel breakdown due to caries with no visible dentine
  4. Underlying dark shadow from dentine
  5. Distinct cavity with visible dentine
  6. Extensive distinct cavity with visible dentine. During the study, a change from level to lower level number (e.g. from 2 to 1) in patients means that the carious lesion is regressed.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 31 | 34
Participants | 9 | 2

4. Secondary Outcome: Caries Activity Assessment According to Nyvad Criteria
Description: Caries activity assessment according to Nyvad criteria, number of participants still have active lesions overall study.
  This assessment includes two clinical judgment inserts: active lesion or inactive lesion basing on visual-tactile surface characteristics of the caries lesions such as integrity, texture, translucency/opacity, lesion location, and surface color.
  During the study, an alteration from active lesion to in active lesion means an improvement.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 31 | 34
Participants | 6 | 21

ADVERSE EVENTS:
Time Frame: 6 months
Description: Incidence of Treatment-Emergent Adverse Events (definitions are adapted from Directive 2001/20/EC and in accordance with ISO 14155 and MDD 93/42). Safety definitions are adapted from the Directive 2001/20/EC and in accordance with ISO 14155 and MDD 93/42.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes